CLINICAL TRIAL: NCT00453752
Title: Non-Invasive Diagnostic and Functional Evaluation of Cardiac Involvement in Patients With Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Other Study IDs: KB/66/2006
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2006-03

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; pulmonary hypertension; echocardiography; N-Terminal proBNP
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study was to assess serum N-terminal proBNP (NT-proBNP) in systemic sclerosis patients and to establish whether it reflects the severity of RV overload.

DETAILED DESCRIPTION:
Elevated serum brain natriuretic peptide (BNP) levels released from myocytes of ventricles upon stretch have been found in patients with isolated right ventricular (RV) pressure overload. However, limited data suggest that serum BNP may be elevated in patients with systemic sclerosis (SSc), especially with RV dysfunction. The aim of this study was to assess serum N-terminal proBNP (NT-proBNP) in SSc patients and to establish whether it reflects the severity of RV overload.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of systemic sclerosis

Exclusion Criteria:

* Cardiovascular disorders other than pulmonary hypertension
* Significant pulmonary function abnormalities
* Impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-04; Study Completion 2010-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michał Ciurzyński, M.D., Ph.D, Principal Investigator — Medical University of Warsaw
Locations (1):
- Michał Ciurzyński, Warsaw, Lindleya 4, Poland